CLINICAL TRIAL: NCT05731310
Title: Efficacy Evaluation and Evaluation of Peripheral Neuroprotective Mechanism of Amgong Niuhuang Pill Combined With Supervised Pulse Music Electroacupuncture on Cognitive Impairment After Ischemic Stroke
Brief Title: Clinical Study of Angong Niuhuang Pill and Acupuncture on PSCI Angong Niuhuang Pill Combined With Supervised Pulse Music Electroacupuncture on Cognitive Impairment After Ischemic Stroke
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0507
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Post-stroke Cognitive Impairment
Keywords: Post-stroke cognitive impairment;acupuncture
MeSH Terms: interventions — Angong Niuhuang Pill

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Angong Niuhuang Pill Group (Experimental): Take half an Angong Niuhuang pill every day for 4 weeks
  Interventions: Drug: Angong Niuhuang Pill
- Angong Niuhuang pill combined with music electroacupuncture group (Experimental): Take half an Angong Niuhuang pill every day for 4 weeks and Daily music scalp acupuncture treatment
  Interventions: Drug: Angong Niuhuang Pill
- General control group (No Intervention): no intervention

INTERVENTIONS:
Drug: Angong Niuhuang Pill — Take Angong Niuhuang pill half a pill/day； Angong Niuhuang pill combined with music scalp acupuncture group These operations last for 4 weeks
  Other Names: Angong Niuhuang pill combined with music scalp acupuncture group
  Arms: Angong Niuhuang Pill Group; Angong Niuhuang pill combined with music electroacupuncture group

SUMMARY:
Post stroke cognitive impairment (PSCI) refers to the attainment of cognitive impairment after the clinical event of stroke A range of syndromes that impede diagnostic criteria. Epidemiologically, PSCI is one of the common complications in stroke patients

DETAILED DESCRIPTION:
(1) Clinical scale data of cognitive function, daily living ability of PSCI patients integrated with the research of this project using uterine Niu Huang pill combined with examined pulse music electroacupuncture

For analysis, the efficacy of PSCI patients was observed; (2) In depth studies on auditory event-related potentials of PSCI treated by uterine Niu Huang pill combined with examined pulse music electroacupuncture

The changes of serum related nerve growth factor and the relationship between each other in order to enrich / fill our province's research results in this field; (3) In key academic journals

1 high level scientific research paper published.

ELIGIBILITY:
Inclusion Criteria:

(1) All were the first stroke, confirmed by head computed tomography (CT) or magnetic resonance imaging (MRI), with vital signs

stable; (2) Those who are conscious and can cooperate with relevant treatment; (3) Montreal Cognitive Assessment Scale (MoCA) score ≤ 24 points; （4）

The course of disease is more than 1 month, and the patient is 40-70 years old.

Exclusion Criteria:

(1) People with cognitive impairment before onset; (2) There are contraindications of Angong Niuhuang Pill or electroacupuncture treatment;

(3) Complicated with dysfunction of heart, liver, kidney and other important organs; (4) Previous history of cerebral hemorrhage, epilepsy, brain injury, etc; (5) Before onset

Have a history of alcohol and drug dependence; (6) The condition worsens, and new hemorrhagic or infarcted foci appear.

-

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Simple intelligence state examination scale | up to 4 weeks
  MMSE

CONTACTS AND LOCATIONS:
Overall Officials: le zhang, Study Chair — 2nd Affiliated Hospital, School of Medicine
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Hangzhou, Zhejiang, China